CLINICAL TRIAL: NCT00930397
Title: The Evaluation of UTERO - Placental 3D Doppler Examination Potential Interest for Pre- Eclampsia Screening During Pregnancy. Observational Study in 100 Women at High Risk for Pre- Eclampsia and 70 Low Risk Women.
Brief Title: Observational Study in UTERO - Placental 3D Doppler Examination: Interest for Pre-eclampsia Screening During Pregnancy
Acronym: PLACENTA3D
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: GE Medical Systems ultrasound (only technical support) (Unknown)
Responsible Party: Sponsor
Other Study IDs: CRC 07049
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2013-05

CONDITIONS: Pre-eclampsia; Intra-uterine Growth Restriction; Placental Insufficiency; 3D Doppler Ultrasound
Keywords: Pre-eclampsia; UTERO-placental unit vascularization; Hypertension, pregnancy- induced; IUGR; Screening; 3D Doppler Ultrasound
MeSH Terms: conditions — Pre-Eclampsia; Placental Insufficiency; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low risk women: Women without any personal risk.
- High risk women: Women at high risk for pre-eclampsia with personal of pre-eclampsia and/or IUGR in a previous pregnancy, diabetes, auto-immune syndrome such as lupus, hypertension, renal insufficiency and anti-phospholipid.

SUMMARY:
Pre-eclampsia and intra uterine growth restriction (IUGR) represent major complications for pregnant women, with a high related maternal and fetal morbidity and mortality. It is now widely admitted that these pathologies, which can concern up to 7% of pregnancies, are in relation with hypo-perfusion of the placenta because of an early deficient trophoblast invasion and uterine vascular remodelling.Advances in ultrasound imaging now permit non invasive 3D volume and Doppler signal quantification using automatic acquisitions.Quantitative comparison of volumes and Doppler parameters between control pregnancies and IUGR ought to confirm the theory of UTERO-placental hypo-perfusion. This technique might allow an earlier prediction for IUGR. The aim of this study is to evaluate the interest of 3D Doppler quantification as a new screening tool for pre eclampsia and IUGR.

DETAILED DESCRIPTION:
One hundred high risk women and 70 low risk women will be included. Inclusion criteria for the high risk group are: personal history of pre eclampsia and/or IUGR in a previous pregnancy, diabetes, auto-immune syndrome such as LUPUS, hypertension, renal insufficiency, and anti-phospholipid syndrome.Patients (over 18 years old) will be included between 11 and 14(+6days) WG. Only singletons pregnancies will be included.3D Doppler standardized acquisitions of the UTERO-placental unit will be performed at each usual ultrasound examination of the pregnancy.Data will be analysed after delivery, in terms of quantified Doppler values, comparing two groups: pregnancies with pre eclampsia / IUGR (group with pathology) and normal pregnancies (control group).This is an observational study.

ELIGIBILITY:
Inclusion Criteria:

* Age eligible for study up to 18 years
* Gestational age between 11 to 14 weeks for the first visit (first-trimester pregnancy).-Singleton pregnancy
* Consent to participate in the study
* Patients affiliated to social security

Group 1:

-Personal History of:

* Preeclampsia during a previous pregnancy: Blood pressure more than 140 mmHg systolic and/or 90 mmHg diastolic + proteinuria
* Diabetes
* IUGR during a previous pregnancy (birth weight < 10th centile)
* Hypertension
* Renal insufficiency
* Autoimmune Disease : Antiphospholipid syndrome

Group 2:Absence of all the Group 1 affiliation criteria.

Exclusion Criteria:

* Participating in the study
* Unability to understand the study
* Set back of patient consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 women high risk of pre-eclampsia and 70 women low risk women of pre-eclampsia
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2009-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Existence of pre eclampsia and/or IUGR | at the end of the pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MOREL, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital LARIBOISIERE Service de gynécologie- obstétrique, Paris, France